CLINICAL TRIAL: NCT01328288
Title: The Thai Pediatric HIV Disease Progression: An Observational Database
Brief Title: Progress Pediatric Study
Status: Completed | Type: Observational
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Bamrasnaradura Infectious Diseases Institute (Other Government); Mahidol University (Other); Chiangrai Prachanukroh Hospital (Other); Sanpatong Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: HIV-NAT 154
Record Dates: First submitted 2011-03-02; First posted 2011-04-04 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: HIV; Depression
Keywords: HIV related adverse events; Immunological failure; virological failure; quality of life; depression; genotypic resistance
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: long-term follow-up of HIV-infected children
  Interventions: Drug: standard ART according to the Thai Ministry of Public Health national guidelines

INTERVENTIONS:
Drug: standard ART according to the Thai Ministry of Public Health national guidelines — Patients may receive any of the standard regimens. These regimens are recommended in the Thai Ministry of Public Health National guidelines for the treatment of HIV in children. Change of treatment will be according to the treating physicians.

SUMMARY:
The purpose of this study is to study the HIV disease progression in HIV-infected Thai children.

DETAILED DESCRIPTION:
This is a multicenter, observational cohort study. HIV-infected children from 5 institutions are followed to assess HIV disease progression: 1. Bamrasnaradura infectious disease institute,2. Faculty of Medicine Siriraj Hospital, Mahidol University, 3. Chiangrai Prachanukroh Hospital, 4. Sanpatong Hospital and 5. HIV-NAT, Thai Red Cross AIDS Research Center.

ELIGIBILITY:
Inclusion Criteria:

1. age < 18 years old
2. Have confirmed HIV infection (ELISA,HIV-DNA PCR,HIV-RNA PCR)
3. Signed consent form

Exclusion Criteria:

1. Hospitalization
2. Emergency case
3. Incomplete Medical Record

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: long-term follow-up of HIV-infected children from: 1. Bamrasnaradura infectious disease institute, 2. Faculty of Medicine Siriraj Hospital, Mahidol University, 3. Chiangrai Prachanukroh Hospital, Chiang Rai, 4. Sanpatong Hospital, Chiang Mai, and 5. HIV-NAT, Thai Red Cross AIDS Research Center, Bangkok
Sampling Method: Probability Sample
Enrollment: 840 (Actual)
Dates: Start 2009-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
HIV related adverse events | 1 year
  time to HIV related adverse events

SECONDARY OUTCOMES:
Immunological failure | 1 year
  time to immunological failure
virological failure | 1 year
  time to virological failure
quality of life | 1 year
  time to change of quality of life
depression | 1 year
  when patient develops depression
genotypic resistance | 1 year
  time to genotypic resistance

CONTACTS AND LOCATIONS:
Overall Officials: Wisit Prasithsirikul, MD, Principal Investigator — Bamrasnaradura infectious disease institute; Rawiwan Hansudewechakul, MD, Principal Investigator — Chiangrai Prachanukroh Hospital; Wirat Klinbuayam, MD, Principal Investigator — Sanpatong Hospital; Jintanat Ananworanich, MD, PhD, Principal Investigator — HIV-NAT, Thai Red Cross - AIDS Research Centre; Kulkanya Chokephaibulkit, MD, Principal Investigator — Mahidol University
Locations (5):
- Thailand (5):
  - Chiangrai Prachanukroh Hospital, Chiang Rai, Changwat Chiang Rai
  - Bamrasnaradura infectious disease institute, Nonthaburi, Changwat Nonthaburi
  - Sanpatong Hospital, Sanpathong, Chiang Mai
  - HIV-NAT, Thai Red Cross AIDS Research Centre, Bangkok
  - Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok

REFERENCES:
- [Result] Bunupuradah T, Sricharoenchai S, Hansudewechakul R, Klinbuayaem V, Teeraananchai S, Wittawatmongkol O, Akarathum N, Prasithsirikul W, Ananworanich J; Pediatric PROGRESS Study Team. Risk of first-line antiretroviral therapy failure in HIV-infected Thai children and adolescents. Pediatr Infect Dis J. 2015 Mar;34(3):e58-62. doi: 10.1097/INF.0000000000000584. PMID 25478649
- See also: HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org